CLINICAL TRIAL: NCT02638259
Title: A Randomized, Double-blind, Parallel-group Phase III Study to Demonstrate Equivalent Efficacy and to Compare Safety & Immunogenicity of GP2015 and Enbrel® (EU Authorized) in Patients With Moderate to Severe, Active Rheumatoid Arthritis
Brief Title: Comparative Efficacy and Safety Study of GP2015 and Enbrel® in Patients With Rheumatoid Arthritis
Acronym: EQUIRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GP15-301
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Biosimilars; Rheumatoid Arthritis; Etanercept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GP2015

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 50mg GP2015 (Experimental): Group 1 will receive treatment with 50mg GP2015 by subcutaneous injection every week up to 24 weeks (Treatment Period 1) after which patients achieving at least a moderate clinical response continue treatment with 50mg GP2015 subcutaneous injection every week up to 48 weeks (Treatment Period 2).
  Interventions: Drug: GP2015
- 50mg EU-authorized Enbrel (Active Comparator): Group 2 will receive treatment with 50mg EU-authorized Enbrel by subcutaneous injection every week up to 24 weeks (Treatment Period 1) after which patients achieving at least a moderate clinical response will be switched to 50 mg GP2015 subcutaneous injection every week up to 48 weeks (Treatment Period 2).
  Interventions: Drug: GP2015

INTERVENTIONS:
Drug: GP2015 — Enbrel comparator

SUMMARY:
Demonstrate equivalent efficacy of GP2015 and EU-authorized Enbrel in patients with moderate to severe, active (RA) who had an inadequate response to disease modifying anti-rheumatic drugs (DMARD) including methotrexate (MTX).

DETAILED DESCRIPTION:
Demonstrate equivalent efficacy of GP2015 and EU-authorized Enbrel in patients with moderate to severe, active (RA) who had an inadequate response to disease modifying anti-rheumatic drugs (DMARD) including methotrexate (MTX). In addition, data on the safety profiles of both products, including immunogenicity and local tolerability at the injection sites, will be collected and compared.

An additional study objective is to identify any potential risk of the transition from Enbrel to GP2015 in terms of general safety and immunogenicity in RA patients

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with RA diagnosis according to ACR 1987 or ACR/EULAR 20110 criteria >/= 6 months at the time of baseline visit
* Patient must have active disease defined as DAS28-CRP>/=3.2
* Patients must have CRP level above ULN >5mg/l) or erythrocyte sedimentation rate (ESR) >/=28mm/h
* Patients must have inadequate clinical response to MTX at a dose of 10-25 mg/wk after proper dose escalation according to local standards

Exclusion Criteria:

* Previous exposure to etanercept in the past
* Patients with functional status class IV according to the ACR 1991 revised criteria
* History of active tuberculosis (TB) or Presence of latent (inactive)TB detected by imaging and/or by the QuantiFERON-TB Gold test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2015-02-21 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2017-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Schwebig, MD, Study Director — Global Program Medical Director
Locations (80):
- United States (24):
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, El Cajon, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Van Nuys, California
  - Novartis Investigative Site, Trumbull, Connecticut
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Zephyrhills, Florida
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Monroe, Louisiana
  - Novartis Investigative Site, Frederick, Maryland
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Orchard Park, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Carrollton, Texas
  - Novartis Investigative Site, Spokane, Washington
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Czechia (4):
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Zlín
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
- Hungary (4):
  - Novartis Investigative Site, Békéscsaba
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szentes
  - Novartis Investigative Site, Szolnok
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rozzano, MI
- Latvia (2):
  - Novartis Investigative Site, Liepāja
  - Novartis Investigative Site, Riga
- Lithuania (4):
  - Novartis Investigative Site, Klaipėda, Klaipėda County
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Panevezys
  - Novartis Investigative Site, Vilnius
- Mexico (4):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Querétaro City
- Poland (6):
  - Novartis Investigative Site, Poznan, Greater Poland Voivodeship
  - Novartis Investigative Site, Lublin, Lublin Voivodeship
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Nadarzyn
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (8):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Belgrade, Serbia
- Slovakia (4):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Rimavská Sobota
  - Novartis Investigative Site, Zvolen
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Córdoba
- United Kingdom (4):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Via CSR

REFERENCES:
- [Derived] Thaci D, Gerdes S, Schulze-Koops H, Allanore Y, Kavanaugh A, Both C, Gattu S, Hachaichi S, Matucci-Cerinic M. Patient-Reported Outcome Measures in Patients with Rheumatoid Arthritis, Psoriasis, or Psoriatic Arthritis Treated with GP2015, an Etanercept Biosimilar: Results from Two Phase III Studies (EGALITY and EQUIRA). Drugs R D. 2025 Jun;25(2):107-115. doi: 10.1007/s40268-025-00507-8. Epub 2025 Apr 25. PMID 40279006
- [Derived] Jaworski J, Matucci-Cerinic M, Schulze-Koops H, Buch MH, Kucharz EJ, Allanore Y, Kavanaugh A, Young P, Babic G. Switch from reference etanercept to SDZ ETN, an etanercept biosimilar, does not impact efficacy, safety, and immunogenicity of etanercept in patients with moderate-to-severe rheumatoid arthritis: 48-week results from the phase III, randomized, double-blind EQUIRA study. Arthritis Res Ther. 2019 May 28;21(1):130. doi: 10.1186/s13075-019-1907-x. PMID 31138316
- [Derived] Matucci-Cerinic M, Allanore Y, Kavanaugh A, Buch MH, Schulze-Koops H, Kucharz EJ, Woehling H, Babic G, Poetzl J, Davis A, Schwebig A. Efficacy, safety and immunogenicity of GP2015, an etanercept biosimilar, compared with the reference etanercept in patients with moderate-to-severe rheumatoid arthritis: 24-week results from the comparative phase III, randomised, double-blind EQUIRA study. RMD Open. 2018 Nov 14;4(2):e000757. doi: 10.1136/rmdopen-2018-000757. eCollection 2018. PMID 30487998

RESULTS

PARTICIPANT FLOW:
Groups:
- 50mg GP2015: Group 1 received treatment with 50mg GP2015 by subcutaneous injection every week up to 24 weeks (Treatment Period 1) after which patients achieving at least a moderate clinical response continued treatment with 50mg GP2015 subcutaneous injection every week up to 48 weeks (Treatment Period 2). GP2015: Enbrel comparator
- 50mg EU-authorized Enbrel: Group 2 will receive treatment with 50mg EU-authorized Enbrel by subcutaneous injection every week up to 24 weeks (Treatment Period 1) after which patients achieving at least a moderate clinical response will be switched to 50 mg GP2015 subcutaneous injection every week up to 48 weeks (Treatment Period 2). GP2015: Enbrel comparator
Period: Treatment Period 1
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Started | 186 | 190
Completed | 181 | 172
Not Completed | 5 | 18
Not completed — Adverse Event | 1 | 5
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Withdrawn per sponsor decision | 0 | 2
Period: Treatment Period 2
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Started | 175 (6 patients did not proceed to TP2 (3 not eligible, 2 consent withdrawal, 1 IP delay)) | 166 (6 patients did not proceed to TP2 (4 not eligible, 1 consent withdrawal, 1 adverse event).)
Completed | 169 | 155
Not Completed | 6 | 11
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 1 | 7

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for Full Analysis Set (FAS). The FAS is comprised of all randomized patients to whom study treatment has been assigned.
Groups:
- 50mg EU-authorized Enbrel: Group 2 received treatment with 50mg EU-authorized Enbrel by subcutaneous injection every week up to 24 weeks (Treatment Period 1) after which patients achieving at least a moderate clinical response were switched to 50 mg GP2015 subcutaneous injection every week up to 48 weeks (Treatment Period 2). GP2015: Enbrel comparator
- Total: Total of all reporting groups
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel | Total
Number analyzed (Participants) | 186 | 190 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.22) | 53.1 (12.70) | 54.1 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 150 | 308
  Male | 28 | 40 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 180 | 185 | 365
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 7 | 12 | 19
  United States | 23 | 26 | 49
  Czechia | 16 | 15 | 31
  United Kingdom | 3 | 4 | 7
  Spain | 5 | 5 | 10
  Russia | 12 | 10 | 22
  Latvia | 6 | 2 | 8
  Poland | 44 | 48 | 92
  Italy | 1 | 0 | 1
  Mexico | 4 | 5 | 9
  Slovakia | 3 | 5 | 8
  Bulgaria | 11 | 11 | 22
  Lithuania | 9 | 12 | 21
  Serbia | 12 | 10 | 22
  Germany | 4 | 5 | 9
  Estonia | 26 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Safety: Change in DAS28-CRP Score From Baseline to Week 24 in Patients Treated With GP2015 and Patients Treated With Enbrel
Description: Disease activity score (DAS) 28-CRP is based on 28-joint count (tender and swollen joints), C-reactive protein and patient's assessment of global disease activity, values range from 0.96 to 10.0 while higher values mean a higher disease activity. • A DAS28-CRP value >5.1 corresponds to a high disease activity • A DAS28-CRP value between 3.2 and 5.1 corresponds to a moderate disease activity • A DAS28-CRP value between 2.6 and 3.2 corresponds to a low disease activity • A DAS28-CRP value < 2.6 corresponds to remission DAS28-CRP = 0.56 * sqrt(tender28) + 0.28* sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * GDA + 0.96 where • tender28 and swollen28 are the number of tender and swollen joints as assessed using 28-joint count • CRP is C-reactive protein (mg/l) • GDA is the global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm
Time Frame: treatment period 1: up to 24 weeks
Population: Treatment Period 1 Per-Protocol set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
scores on a scale | -2.80 (0.113) | -2.73 (0.117)
Statistical Analysis 1: Comparison: 50mg GP2015 vs 50mg EU-authorized Enbrel; Therapeutic equivalence in terms of change from baseline in DAS28-CRP at week 24 will be concluded if the 95% confidence interval for the LS mean difference between GP2015 and Enbrel is contained within the interval [-0.6; 0.6]. A mixed-model repeated measures analysis was performed for DAS28-CRP change from baseline including treatment, stratification factors, time, the interaction between time (visits) and treatment all as categorical variables, and baseline DAS28-CRP as a continuous variable; Test type: Equivalence — A margin of 0.6 can be statistically and clinically justified based on the results Keystone et al, Arthritis and Rheumatism, p353-363, (2004) and on the EULAR response criteria. The sample size of 155 per group with 90% power is based on the common SD of 1.46 and was calculated using nQuery 7.0; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.26 to 0.12], Standard Error of Mean 0.097

2. Secondary Outcome: Treatment Period 1: Frequency and Severity of Injection Site Reactions in GP2015 and Enbrel
Description: Frequency of participants with injection site reactions in GP2015 and Enbrel
Time Frame: Treatment Period 1, up to 24 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 186 | 190
Participants
  All injection site reactions | 13 | 35
  Moderate injection site reactions | 1 | 5
  Severe injection site reactions | 0 | 0

3. Secondary Outcome: Treatment Period 1 - Safety : Immunogenicity by Measuring the Rate of Anti-drug Antibody (ADA) Positive Patients
Description: Frequency of patients having anti-drug antibody (ADA) during 24 weeks (Treatment Period 1) using 1% false positive rate
Time Frame: baseline, week 2, week 4, week 12, week 24
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 186 | 190
Participants
  Baseline | 2 | 0
  Week 2 | 2 | 5
  Week 4 | 3 | 42
  Week 12 | 0 | 5
  Week 24 | 0 | 0

4. Secondary Outcome: Treatment Period 1- DAS28-CRP and DAS28-erythrocyte Sedimentation Rate (ESR) Scores at Baseline and Weeks 4, 12 and 24;
Description: DAS28-CRP is a disease activity score and defined in primary outcome measure. DAS28-ESR is the DAS28 erythrocyte sedimentation rate score.
  DAS28-CRP and DAS28-ESR:
  1. best is 0,
  2. < 2.6 - remission,
  3. ≥ 2.6 to ≤ 3.2 - low disease activity
  4. > 3.2 to ≤ 5.1 - moderate disease activity
  5. > 5.1 - high disease activity
  DAS28-ESR = 0.56 * sqrt(tender28) + 0.28* sqrt(swollen28) + 0.7 * ln(ESR) + 0.014 * GDA where • tender28 and swollen28 are the number of tender and swollen joints as assessed using 28-joint count • CRP is C-reactive protein (mg/l) • ESR is erythrocyte sedimentation rate (mm/h) • GDA is the global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm
Time Frame: week 4, 12, 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
score on a scale
  DAS28-CRP baseline | 5.42 (0.921) | 5.53 (0.783)
  DAS28-CRP week 4: number analyzed (Participants) | 165 | 153
  DAS28-CRP week 4 | 3.81 (1.079) | 3.82 (1.077)
  DAS28-CRP week 12: number analyzed (Participants) | 165 | 150
  DAS28-CRP week 12 | 3.15 (1.045) | 3.31 (1.088)
  DAS28-CRP week 24 | 2.63 (0.910) | 2.75 (0.928)
  DAS28-ESR baseline | 6.34 (0.882) | 6.41 (0.768)
  DAS28-ESR week 4: number analyzed (Participants) | 167 | 154
  DAS28-ESR week 4 | 4.62 (1.183) | 4.56 (1.204)
  DAS28-ESR week 12: number analyzed (Participants) | 168 | 154
  DAS28-ESR week 12 | 3.84 (1.216) | 3.94 (1.284)
  DAS28-ESR week 24 | 3.24 (1.060) | 3.32 (1.099)

5. Secondary Outcome: Treatment Period 1 - Changes From Baseline in DAS28-CRP and DAS-ESR Scores to Weeks 4, 12 and 24
Time Frame: baseline, Week 4, week 12, week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
score on a scale
  DAS28-CRP change from baseline week 4: number analyzed (Participants) | 165 | 153
  DAS28-CRP change from baseline week 4 | -1.59 (1.032) | -1.70 (1.001)
  DAS28-CRP change from baseline week 12: number analyzed (Participants) | 165 | 150
  DAS28-CRP change from baseline week 12 | -2.23 (1.030) | -2.20 (1.071)
  DAS28-CRP change from baseline week 24 | -2.78 (1.058) | -2.78 (1.028)
  DAS28-ESR change from baseline week 4: number analyzed (Participants) | 167 | 154
  DAS28-ESR change from baseline week 4 | -1.72 (1.068) | -1.85 (1.078)
  DAS28-ESR change from baseline week 12: number analyzed (Participants) | 168 | 154
  DAS28-ESR change from baseline week 12 | -2.50 (1.145) | -2.47 (1.218)
  DAS28-ESR change from baseline week 24 | -3.10 (1.157) | -3.09 (1.119)

6. Secondary Outcome: Treatment Period 1- Proportion of Patients Achieving EULAR Response
Description: Proportion of patients achieving European League against Rheumatism (EULAR) good response (defined as DAS28 ≤ 3.2 and DAS28 improvement from Baseline > 1.2) and moderate response (defined as DAS28 ≤ 3.2 and DAS28 improvement > 0.6 and ≤ 1.2, or DAS28 > 3.2 and ≤ 5.1 and DAS28 improvement > 0.6 or DAS28 > 5.1 but DAS28 improvement > 1.2) ;
Time Frame: week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  Good response week 4: number analyzed (Participants) | 167 | 154
  Good response week 4 | 26 | 21
  Good response week 12: number analyzed (Participants) | 168 | 154
  Good response week 12 | 54 | 47
  Good response week 24 | 88 | 74
  Moderate response week 4: number analyzed (Participants) | 167 | 154
  Moderate response week 4 | 95 | 99
  Moderate response week 12: number analyzed (Participants) | 168 | 154
  Moderate response week 12 | 103 | 91
  Moderate response week 24 | 76 | 77
  no response week 4: number analyzed (Participants) | 167 | 154
  no response week 4 | 46 | 34
  no response week 12: number analyzed (Participants) | 168 | 154
  no response week 12 | 11 | 16
  no response week 24 | 4 | 4

7. Secondary Outcome: Treatment Period 1- Proportion of Patients Achieving DAS28 < 2.6 at Weeks 4, 12 and 24
Description: % patients in DAS28-ESR categories up to week 24
Time Frame: week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  Week 4 - remission (DAS28 <2.6) | 9 | 7
  Week 12 - remission (DAS28 <2.6) | 21 | 21
  Week 24 - remission (DAS28 <2.6) | 46 | 41

8. Secondary Outcome: Treatment Period 1- Proportion of Patients Achieving EULAR/ACR Boolean Remission Criteria
Description: Proportion of patients achieving EULAR/American College of Rheumatology (EULAR/ACR) Boolean remission criteria (defined as number of tender joints/swollen joints ≤ 1 and CRP (mg/dL) ≤ 1 and patient global assessment (1-10) ≤ 1) at Weeks 4, 12 and 24;
Time Frame: week 4, week 12, week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  week 4: number analyzed (Participants) | 165 | 153
  week 4 | 1 | 2
  week 12: number analyzed (Participants) | 165 | 150
  week 12 | 9 | 8
  week 24 | 24 | 15

9. Secondary Outcome: Treatment Period 1- Proportion of Patients Achieving ACR20/50/70 Response at Weeks 4, 12 and 24;
Description: ACR20 response was defined if a patient fulfilled all 3 criteria below:
  * 20% improvement in tender 68 joint-count
  * 20% improvement in swollen 68 joint-count;
  And 20% improvement in at least 3 of the following 5 measures:
  * Patient's assessment of RA pain (visual analogue scale (VAS) 100 mm),
  * Patient's global assessment of disease activity (VAS 100 mm),
  * Physician's global assessment of disease activity (VAS 100 mm),
  * Patient self-assessed disability (HAQ score),
  * Acute phase reactant (CRP or ESR). ACR50 and ACR70 responses were defined as ACR20 response replacing "20% improvement" by "50% improvement" and "70% improvement", respectively.
Time Frame: Week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  ACR20 response Week 4: number analyzed (Participants) | 166 | 154
  ACR20 response Week 4 | 80 | 83
  ACR20 response Week 12: number analyzed (Participants) | 166 | 154
  ACR20 response Week 12 | 131 | 116
  ACR20 response Week 24: number analyzed (Participants) | 167 | 155
  ACR20 response Week 24 | 147 | 144
  ACR50 response Week 4: number analyzed (Participants) | 166 | 154
  ACR50 response Week 4 | 25 | 28
  ACR50 response Week 12: number analyzed (Participants) | 166 | 154
  ACR50 response Week 12 | 55 | 68
  ACR50 response Week 24: number analyzed (Participants) | 167 | 155
  ACR50 response Week 24 | 107 | 110
  ACR70 response Week 4: number analyzed (Participants) | 166 | 154
  ACR70 response Week 4 | 8 | 7
  ACR70 response Week 12: number analyzed (Participants) | 166 | 154
  ACR70 response Week 12 | 21 | 26
  ACR70 response Week 24: number analyzed (Participants) | 167 | 155
  ACR70 response Week 24 | 56 | 66

10. Secondary Outcome: Treatment Period 1- ACR-N Scores at Weeks 4, 12 and 24;
Description: ACR-N (American College of Rheumatology percentage of improvement): negative is worsening, positive (up to 100) is an improvement.
  ACR-N is a single number that characterizes the percentage of improvement from Baseline that a patient has experienced in analogy to ACR20 described above. ACR-N of X (such as 38) means that the patient had achieved an improvement of at least X% (such as 38%) in tender and swollen joints, and an improvement of at least X% (such as 38%) in 3 of the 5 other parameters mentioned above.
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
score on a scale
  week 4: number analyzed (Participants) | 166 | 154
  week 4 | 19.9 (29.89) | 22.6 (34.02)
  week 12: number analyzed (Participants) | 166 | 154
  week 12 | 38.3 (27.46) | 38.7 (35.32)
  week 24: number analyzed (Participants) | 167 | 155
  week 24 | 55.4 (27.61) | 59.4 (25.40)

11. Secondary Outcome: Treatment Period 1 - Proportion of Patients in Each Disease Activity Category as Defined by SDAI
Description: Proportion of patients in each disease activity category as defined by the Simplified Disease Activity Index (SDAI): high disease activity, SDAI > 26, moderate disease activity, SDAI > 11 to ≤ 26, low disease activity, SDAI > 3.3 to ≤ 11, and remission, SDAI ≤ 3.3 at Weeks 4, 12 and 24; SDAI and CDAI are measures of disease activity in RA. The scores were calculated by numerical summation of the number of tender and swollen joints (using the 28-joint count), and the patient's and physician's global assessment of disease activity.
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  Baseline : Remission (SDAI<=3.3) | 0 | 0
  Baseline: Low (3.3 < SDAI <= 11) | 0 | 0
  Baseline : Moderate (11 < SDAI <= 26 | 26 | 19
  Baseline : High (SDAI > 26) | 142 | 136
  Week 4:Remission (SDAI<=3.3) | 5 | 4
  Week 4:Low (3.3 < SDAI <= 11) | 35 | 31
  Week 4: Moderate (11 < SDAI <= 26 | 84 | 82
  Week 4:High (SDAI > 26) | 41 | 36
  Week 12:Remission (SDAI<=3.3) | 15 | 13
  Week 12:Low (3.3 < SDAI <= 11) | 61 | 58
  Week 12: Moderate (11 < SDAI <= 26 | 75 | 68
  Week 12:High (SDAI > 26) | 14 | 11
  Week 24: Remission (SDAI<=3.3) | 38 | 31
  Week 24: Low (3.3 < SDAI <= 11) | 83 | 81
  Week 24 : Moderate (11 < SDAI <= 26 | 45 | 38
  Week 24 :High (SDAI > 26) | 2 | 5

12. Secondary Outcome: Treatment Period 1 - Proportion of Patients in Each Disease Activity Category as Defined by CDAI
Description: Proportion of patients in each disease activity category as defined by the Clinical Disease Activity Index (CDAI): high disease activity, CDAI > 22, moderate disease activity, CDAI > 10 to ≤ 22, low disease activity, CDAI > 2.8 to ≤ 10, and remission, CDAI ≤ 2.8 at Weeks 4, 12 and 24; SDAI and CDAI are measures of disease activity in RA. The scores were calculated by numerical summation of the number of tender and swollen joints (using the 28-joint count), and the patient's and physician's global assessment of disease activity.
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  Baseline : Remission (CDAI<=2.8) | 0 | 0
  Baseline: Low (2.8 < CDAI <= 10) | 0 | 0
  Baseline : Moderate (10 < CDAI <= 22 | 17 | 7
  Baseline : High (CDAI > 22) | 151 | 148
  Week 4:Remission(CDAI<=2.8) | 4 | 3
  Week 4: Low (2.8 < CDAI <= 10) | 33 | 31
  Week 4: Moderate (10 < CDAI <= 22) | 67 | 71
  Week 4:High High (CDAI > 22) | 63 | 49
  Week 12:Remission(CDAI<=2.8) | 14 | 15
  Week 12: Low (2.8 < CDAI <= 10) | 63 | 53
  Week 12: Moderate (10 < CDAI <= 22) | 72 | 63
  Week 12:High (CDAI > 22) | 19 | 23
  Week 24: Remission (CDAI<=2.8) | 35 | 31
  Week 24: Low (2.8 < CDAI <= 10) | 81 | 78
  Week 24 : (10 < CDAI <= 22) | 46 | 39
  Week 24 :High (CDAI > 22) | 6 | 7

13. Secondary Outcome: Treatment Period 1- Proportion of Patients Achieving HAQ Index in Normal Range (≤ 0.5) at Weeks 4, 12 and 24;
Description: Health assessment questionnaire (HAQ) disability index ranges from 0 (best) to 3 (worst)
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
Participants
  Baseline: number analyzed (Participants) | 168 | 154
  Baseline | 11 | 5
  Week 4: number analyzed (Participants) | 167 | 153
  Week 4 | 22 | 30
  Week 12: number analyzed (Participants) | 168 | 154
  Week 12 | 40 | 46
  Week 24: number analyzed (Participants) | 166 | 152
  Week 24 | 54 | 62

14. Secondary Outcome: Treatment Period 1 - Health Assessment Questionnaire (HAQ) Index at Baseline, Weeks 4, 12 and 24;
Description: Health assessment questionnaire (HAQ) disability index ranges from 0 (best) to 3 (worst)
Time Frame: Baseline, Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
score on a scale
  Baseline | 1.44 (0.547) | 1.47 (0.561)
  Week 4: number analyzed (Participants) | 167 | 153
  Week 4 | 1.19 (0.558) | 1.14 (0.611)
  Week 12: number analyzed (Participants) | 168 | 154
  Week 12 | 1.02 (0.560) | 0.97 (0.599)
  Week 24: number analyzed (Participants) | 166 | 152
  Week 24 | 0.88 (0.601) | 0.80 (0.589)

15. Secondary Outcome: Treatment Period 1 - Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale Relative to Baseline at Weeks 4, 12 and 24;
Description: FACIT fatigue scale is a 13- item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function, ranging from 0 (worst) to 52 (best). A score of less than 30 indicates severe fatigue.
Time Frame: Baseline, Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
score on a scale
  Baseline: number analyzed (Participants) | 156 | 146
  Baseline | 27.0 (9.67) | 25.1 (10.33)
  Week 4: number analyzed (Participants) | 167 | 154
  Week 4 | 31.6 (8.83) | 30.9 (10.01)
  Week 12: number analyzed (Participants) | 168 | 154
  Week 12 | 34.4 (8.93) | 33.9 (9.6)
  Week 24 | 36.3 (8.94) | 36.7 (9.24)

16. Secondary Outcome: Treatment Period 1 - CRP Levels at Baseline and Weeks 4, 12 and 24
Time Frame: Weeks 4, 12 and 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
mg/dL
  Baseline | 1.19 (2.194) | 1.10 (1.526)
  Week 4: number analyzed (Participants) | 165 | 153
  Week 4 | 0.36 (0.718) | 0.43 (0.693)
  Week 12: number analyzed (Participants) | 165 | 150
  Week 12 | 0.33 (0.772) | 0.48 (0.850)
  Week 24 | 0.44 (0.949) | 0.35 (0.466)

17. Secondary Outcome: Treatment Period 1 - ESR Levels at Baseline and Weeks 4, 12 and 24
Time Frame: Weeks 4, 12 and 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 168 | 155
mm/h
  Baseline | 41.4 (16.89) | 41.8 (17.94)
  Week 4: number analyzed (Participants) | 167 | 154
  Week 4 | 26.5 (16.51) | 26.7 (17.27)
  Week 12: number analyzed (Participants) | 168 | 154
  Week 12 | 23.2 (14.67) | 23.8 (15.41)
  Week 24 | 21.4 (15.47) | 20.8 (14.05)

18. Secondary Outcome: Treatment Period 2: DAS28-CRP and DAS28-ESR Scores up to Week 48;
Description: DAS28-CRP and DAS28-ESR:
  1. best is 0,
  2. < 2.6 - remission,
  3. ≥ 2.6 to ≤ 3.2 - low disease activity
  4. > 3.2 to ≤ 5.1 - moderate disease activity
  5. > 5.1 - high disease activity
Time Frame: Baseline, week 4, week 12, week 24, week 36 and week 48.
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
score on a scale
  DAS28-CRP Baseline | 5.45 (0.914) | 5.57 (0.794)
  DAS28-CRP Week 4: number analyzed (Participants) | 145 | 129
  DAS28-CRP Week 4 | 3.89 (1.053) | 3.79 (1.101)
  DAS28-CRP Week 12: number analyzed (Participants) | 146 | 127
  DAS28-CRP Week 12 | 3.20 (1.038) | 3.27 (1.127)
  DAS28-CRP Week 24 | 2.64 (0.863) | 2.67 (0.892)
  DAS28-CRP Week 36: number analyzed (Participants) | 147 | 130
  DAS28-CRP Week 36 | 2.65 (1.001) | 2.74 (1.017)
  DAS28-CRP Week 48 | 2.57 (1.067) | 2.74 (1.062)
  DAS28-ESR Baseline | 6.39 (0.872) | 6.43 (0.784)
  DAS28-ESR Week 4: number analyzed (Participants) | 147 | 130
  DAS28-ESR Week 4 | 4.70 (1.175) | 4.49 (1.228)
  DAS28-ESR Week 12: number analyzed (Participants) | 148 | 130
  DAS28-ESR Week 12 | 3.90 (1.236) | 3.85 (1.317)
  DAS28-ESR Week 24 | 3.23 (1.022) | 3.19 (1.048)
  DAS28-ESR Week 36: number analyzed (Participants) | 147 | 131
  DAS28-ESR Week 36 | 3.25 (1.160) | 3.28 (1.127)
  DAS28-ESR Week 48: number analyzed (Participants) | 147 | 129
  DAS28-ESR Week 48 | 3.20 (1.201) | 3.30 (1.177)

19. Secondary Outcome: Treatment Period 2 : Changes From Baseline in DAS28-CRP and DAS28-ESR Scores From Week 4 up to Week 48
Time Frame: week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
score on a scale
  DAS28-CRP change from baseline, week 4: number analyzed (Participants) | 145 | 129
  DAS28-CRP change from baseline, week 4 | -1.55 (1.014) | -1.76 (1.014)
  DAS28-CRP change from baseline, week 12: number analyzed (Participants) | 146 | 127
  DAS28-CRP change from baseline, week 12 | -2.22 (1.031) | -2.27 (1.096)
  DAS28-CRP change from baseline, week 24 | -2.81 (1.007) | -2.90 (0.988)
  DAS28-CRP change from baseline, week 36: number analyzed (Participants) | 147 | 130
  DAS28-CRP change from baseline, week 36 | -2.80 (1.087) | -2.82 (1.151)
  DAS28-CRP change from baseline, week 48 | -2.88 (1.198) | -2.83 (1.176)
  DAS28-ESR change from baseline, week 4: number analyzed (Participants) | 147 | 130
  DAS28-ESR change from baseline, week 4 | -1.69 (1.048) | -1.92 (1.087)
  DAS28-ESR change from baseline, week 12: number analyzed (Participants) | 148 | 130
  DAS28-ESR change from baseline, week 12 | -2.49 (1.152) | -2.57 (1.235)
  DAS28-ESR change from baseline, week 24 | -3.16 (1.106) | -3.23 (1.054)
  DAS28-ESR change from baseline, week 36: number analyzed (Participants) | 147 | 131
  DAS28-ESR change from baseline, week 36 | -3.13 (1.232) | -3.14 (1.154)
  DAS28-ESR change from baseline, week 48: number analyzed (Participants) | 147 | 129
  DAS28-ESR change from baseline, week 48 | -3.20 (1.297) | -3.14 (1.190)

20. Secondary Outcome: Treatment Period 2: Proportion of Patients Achieving EULAR Reponse
Description: Proportion of patients achieving EULAR good response (defined as DAS28 ≤ 3.2 and DAS28 improvement from Baseline > 1.2) and moderate response (defined as DAS28 ≤ 3.2 and DAS28 improvement > 0.6 and ≤ 1.2, or DAS28 > 3.2 and ≤ 5.1 and DAS28 improvement > 0.6 or DAS28 > 5.1 but DAS28 improvement > 1.2) at Weeks 36 and 48;
Time Frame: week 4, week 12, week 24, week 36 and week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  Good response week 4: number analyzed (Participants) | 147 | 130
  Good response week 4 | 20 | 20
  Good response week 12: number analyzed (Participants) | 148 | 130
  Good response week 12 | 43 | 43
  Good response week 24 | 77 | 68
  Good response week 36: number analyzed (Participants) | 147 | 131
  Good response week 36 | 82 | 65
  Good response week 48: number analyzed (Participants) | 147 | 129
  Good response week 48 | 80 | 67
  Moderate response week 4: number analyzed (Participants) | 147 | 130
  Moderate response week 4 | 85 | 82
  Moderate response week 12: number analyzed (Participants) | 148 | 130
  Moderate response week 12 | 95 | 75
  Moderate response week 24 | 71 | 63
  Moderate response week 36: number analyzed (Participants) | 147 | 131
  Moderate response week 36 | 62 | 64
  Moderate response week 48: number analyzed (Participants) | 147 | 129
  Moderate response week 48 | 61 | 57
  no response week 4: number analyzed (Participants) | 148 | 130
  no response week 4 | 42 | 28
  no response week 12: number analyzed (Participants) | 148 | 130
  no response week 12 | 10 | 12
  no response week 24 | 0 | 0
  no response week 36: number analyzed (Participants) | 147 | 131
  no response week 36 | 3 | 2
  no response week 48: number analyzed (Participants) | 147 | 129
  no response week 48 | 6 | 5

21. Secondary Outcome: Treatment Period 2 : Proportion of Patients Achieving DAS28 < 2.6 at Weeks 36 and 48;
Description: percentage of participants in DAS28-ESR categories up to week 48
Time Frame: week 36 and week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  Week 36 Remission (DAS28 < 2.6) | 45 | 38
  Week 48 Remission (DAS28 < 2.6) | 44 | 35

22. Secondary Outcome: Treatment Period 2 : Proportion of Patients Achieving EULAR/ACR Boolean Remission Criteria
Description: Proportion of patients achieving EULAR/ACR Boolean remission criteria (defined as number of tender joints/swollen joints ≤ 1 and CRP (mg/dL) ≤ 1 and patient global assessment (1-10) ≤ 1) at Weeks 36 and 48;
Time Frame: week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  Week 4: number analyzed (Participants) | 145 | 129
  Week 4 | 0 | 2
  Week 12: number analyzed (Participants) | 146 | 127
  Week 12 | 9 | 8
  Week 24 | 22 | 13
  Week 36: number analyzed (Participants) | 147 | 130
  Week 36 | 25 | 15
  Week 48 | 28 | 20

23. Secondary Outcome: Treatment Period 2 : Proportion of Patients Achieving ACR20/50/70 Response at Weeks 36 and 48;
Time Frame: week 36 and week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  ACR20 response Week 36: number analyzed (Participants) | 146 | 131
  ACR20 response Week 36 | 128 | 114
  ACR20 response Week 48: number analyzed (Participants) | 147 | 131
  ACR20 response Week 48 | 131 | 108
  ACR50 response Week 36: number analyzed (Participants) | 146 | 131
  ACR50 response Week 36 | 90 | 83
  ACR50 response Week 48: number analyzed (Participants) | 147 | 131
  ACR50 response Week 48 | 93 | 86
  ACR70 response Week 36: number analyzed (Participants) | 146 | 131
  ACR70 response Week 36 | 47 | 50
  ACR70 response Week 48: number analyzed (Participants) | 147 | 131
  ACR70 response Week 48 | 54 | 55

24. Secondary Outcome: Treatment Period 2 : ACR-N Scores at Weeks 36 and 48;
Description: ACR-N: negative is worsening, positive (up to 100) is an improvement
Time Frame: week 36 and week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
score on a scale
  Week 4: number analyzed (Participants) | 146 | 130
  Week 4 | 19.7 (27.72) | 24.9 (29.40)
  Week 12: number analyzed (Participants) | 146 | 130
  Week 12 | 38.3 (27.84) | 40.7 (34.80)
  Week 24: number analyzed (Participants) | 147 | 131
  Week 24 | 56.3 (26.58) | 60.9 (24.79)
  Week 36: number analyzed (Participants) | 146 | 131
  Week 36 | 53.8 (28.21) | 55.7 (28.37)
  Week 48: number analyzed (Participants) | 147 | 131
  Week 48 | 56.9 (29.18) | 56.4 (30.58)

25. Secondary Outcome: Treatment Period 2 : Proportion of Patients in Each Disease Activity Category as Defined by SDAI
Description: Proportion of patients in each disease activity category as defined by the Simplified Disease Activity Index (SDAI): high disease activity, SDAI > 26, moderate disease activity, SDAI > 11 to ≤ 26, low disease activity, SDAI > 3.3 to ≤ 11, and remission, SDAI ≤ 3.3 at Weeks 36 and 48.
Time Frame: baseline, week 4, week 12, week 24, week 36. week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  Baseline : Remission (SDAI <= 3.3) | 0 | 0
  Baseline : Low (3.3 < SDAI <= 11) | 0 | 0
  Baseline : Moderate (11 < SDAI <= 26) | 20 | 16
  Baseline : High (SDAI > 26 ) | 128 | 115
  Week 4 : Remission (SDAI <= 3.3) | 2 | 4
  Week 4 : Low (3.3 < SDAI <= 11) | 29 | 27
  Week 4 : Moderate (11 < SDAI <= 26 | 75 | 69
  Week 4 : High (SDAI > 26 ) | 39 | 29
  Week 12: Remission (SDAI <= 3.3) | 14 | 12
  Week 12 : Low (3.3 < SDAI <= 11) | 50 | 51
  Week 12 : Moderate (11 < SDAI <= 26 | 69 | 53
  Week 12 : High (SDAI > 26 ) | 13 | 11
  Week 24: Remission (SDAI <= 3.3) | 31 | 29
  Week 24 : Low (3.3 < SDAI <= 11) | 74 | 71
  Week 24 : Moderate (11 < SDAI <= 26 | 43 | 29
  Week 24 : High (SDAI > 26 ) | 0 | 2
  Week 36: Remission (SDAI <= 3.3) | 34 | 29
  Week 36 : Low (3.3 < SDAI <= 11 | 69 | 66
  Week 36 : Moderate (11 < SDAI <= 26 | 43 | 30
  Week 36 : High (SDAI > 26 ) | 1 | 5
  Week 48: Remission (SDAI <= 3.3) | 39 | 32
  Week 48 : Low (3.3 < SDAI <= 11 | 72 | 62
  Week 48 : Moderate (11 < SDAI <= 26 | 30 | 29
  Week 48 : High (SDAI > 26 ) | 6 | 8

26. Secondary Outcome: Treatment Period 2 : Proportion of Patients in Each Disease Activity Category as Defined by CDAI
Description: Proportion of patients in each disease activity category as defined by the Clinical Disease Activity Index (CDAI): high disease activity, CDAI > 22, moderate disease activity, CDAI > 10 to ≤ 22, low disease activity, CDAI > 2.8 to ≤ 10, and remission, CDAI ≤ 2.8 at Weeks 36 and 48;
Time Frame: baseline, week 4, week 12, week 24, week 36 and week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  Baseline : Remission (CDAI <=2.8) | 0 | 0
  Baseline : Low (2.8 < CDAI <= 10) | 0 | 0
  Baseline : Moderate (10 < CDAI <= 22) | 14 | 6
  Baseline : High (CDAI > 22 ) | 134 | 125
  Week 4 : Remission (CDAI <=2.8) | 2 | 3
  Week 4 : Low (2.8 < CDAI <= 10) | 27 | 28
  Week 4 : Moderate (11 < SDAI <= 26 | 60 | 60
  Week 4 : High (CDAI > 22 ) | 58 | 39
  Week 12: Remission (CDAI <=2.8) | 12 | 14
  Week 12 : Low (2.8 < CDAI <= 10) | 52 | 47
  Week 12 : Moderate (10 < CDAI <= 22) | 67 | 50
  Week 12 : High (CDAI > 22 ) | 17 | 19
  Week 24: Remission (CDAI <=2.8) | 29 | 29
  Week 24 : Low (2.8 < CDAI <= 10) | 71 | 68
  Week 24 : Moderate (10 < CDAI <= 22) | 45 | 30
  Week 24 : High (CDAI > 22 ) | 3 | 4
  Week 36: Remission (CDAI <=2.8) | 32 | 29
  Week 36 : Low (2.8 < CDAI <= 10) | 67 | 63
  Week 36 : Moderate (10 < CDAI <= 22) | 41 | 32
  Week 36 : High (CDAI > 22 ) | 7 | 7
  Week 48: Remission (CDAI <=2.8) | 37 | 29
  Week 48 : Low (2.8 < CDAI <= 10) | 71 | 63
  Week 48 : Moderate (10 < CDAI <= 22) | 32 | 31
  Week 48 : High (CDAI > 22 ) | 7 | 8

27. Secondary Outcome: Treatment Period 2 :Proportion of Patients Achieving HAQ Index in Normal Range (≤ 0.5) at Weeks 36 and 48;
Time Frame: baseline, week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
Participants
  Baseline: number analyzed (Participants) | 148 | 130
  Baseline | 8 | 4
  Week 4: number analyzed (Participants) | 147 | 129
  Week 4 | 17 | 25
  Week 12: number analyzed (Participants) | 148 | 130
  Week 12 | 33 | 39
  Week 24: number analyzed (Participants) | 147 | 128
  Week 24 | 47 | 51
  Week 36: number analyzed (Participants) | 147 | 130
  Week 36 | 46 | 48
  Week 48: number analyzed (Participants) | 147 | 129
  Week 48 | 51 | 51

28. Secondary Outcome: Treatment Period 2 :HAQ Index at Weeks 36 and 48;
Description: HAQ: from 0 (best) to 3 (worst)
Time Frame: baseline, week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
score on a scale
  Baseline: number analyzed (Participants) | 148 | 129
  Baseline | 1.47 (0.547) | 1.50 (0.554)
  Week 4: number analyzed (Participants) | 147 | 129
  Week 4 | 1.22 (0.554) | 1.14 (0.620)
  Week 12: number analyzed (Participants) | 148 | 127
  Week 12 | 1.04 (0.560) | 0.97 (0.614)
  Week 24: number analyzed (Participants) | 147 | 131
  Week 24 | 0.88 (0.594) | 0.83 (0.603)
  Week 36: number analyzed (Participants) | 147 | 130
  Week 36 | 0.89 (0.584) | 0.85 (0.651)
  Week 48: number analyzed (Participants) | 147 | 129
  Week 48 | 0.85 (0.609) | 0.84 (0.652)

29. Secondary Outcome: Treatment Period 2 : Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale Relative to Baseline at Weeks 36 and 48;
Description: FACIT: from 0 (worst) to 52 (best), a score of less than 30 indicates severe fatigue
Time Frame: baseline, week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
score on a scale
  Baseline: number analyzed (Participants) | 138 | 123
  Baseline | 26.6 (9.71) | 25.5 (10.78)
  Week 4: number analyzed (Participants) | 147 | 130
  Week 4 | 31.5 (8.72) | 31.3 (10.07)
  Week 12: number analyzed (Participants) | 148 | 130
  Week 12 | 34.4 (8.89) | 34.1 (9.69)
  Week 24 | 36.6 (8.75) | 36.7 (9.05)
  Week 36: number analyzed (Participants) | 147 | 131
  Week 36 | 36.9 (8.79) | 36.4 (9.50)
  Week 48 | 38.0 (8.74) | 35.8 (9.97)

30. Secondary Outcome: Treatment Period 2 : CRP Levels at Week 36 and 48
Time Frame: baseline, week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
mg/dL
  Baseline | 1.21 (2.244) | 1.17 (1.589)
  Week 4: number analyzed (Participants) | 145 | 129
  Week 4 | 0.36 (0.733) | 0.42 (0.625)
  Week 12: number analyzed (Participants) | 146 | 127
  Week 12 | 0.36 (0.817) | 0.50 (0.910)
  Week 24 | 0.44 (0.964) | 0.36 (0.487)
  Week 36: number analyzed (Participants) | 146 | 130
  Week 36 | 0.39 (0.758) | 0.39 (0.655)
  Week 48 | 0.35 (0.623) | 0.40 (0.878)

31. Secondary Outcome: Treatment Period 2 : ESR Levels at Week 36 and 48
Time Frame: baseline, week 4, week 12, week 24, week 36, week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 148 | 131
mm/h
  Baseline | 42.2 (16.99) | 41.7 (17.99)
  Week 4: number analyzed (Participants) | 147 | 130
  Week 4 | 26.8 (16.33) | 25.3 (16.11)
  Week 12: number analyzed (Participants) | 148 | 130
  Week 12 | 23.8 (15.07) | 23.0 (15.38)
  Week 24 | 21.3 (15.66) | 19.3 (12.66)
  Week 36: number analyzed (Participants) | 147 | 131
  Week 36 | 22.1 (16.41) | 20.3 (14.28)
  Week 48: number analyzed (Participants) | 147 | 129
  Week 48 | 22.8 (16.66) | 20.8 (14.62)

32. Secondary Outcome: Safety - Overall Study : Frequency and Severity of Injection Site Reactions in GP2015 and Enbrel
Description: Frequency of participants with injection site reactions in GP2015 and Enbrel
Time Frame: up to 48 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 186 | 190
Participants
  participants with at least one ISR | 13 | 37
  participants with at least one moderate ISR | 1 | 7
  participants with at least one severe ISR | 0 | 0

33. Secondary Outcome: Safety : Overall Study: Immunogenicity by Measuring the Rate of Anti-drug Antibody (ADA) Positive Patients
Description: To assess the immunogenicity of continuous GP2015 treatment versus a treatment transition from Enbrel to GP2015 after 24 weeks of treatment by measuring the rate of ADA positive participants at Weeks 24, 30, 36 and 48. summary of ADA positive data up to week 48 using a 1% false positive cut point
Time Frame: baseline, week 4, week 12, week 24, week 36, week 48
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg GP2015 | 50mg EU-authorized Enbrel
Number analyzed (Participants) | 186 | 190
Participants
  Baseline | 2 | 0
  Week 2: number analyzed (Participants) | 183 | 185
  Week 2 | 2 | 5
  Week 4: number analyzed (Participants) | 183 | 185
  Week 4 | 3 | 42
  Week 12: number analyzed (Participants) | 179 | 176
  Week 12 | 0 | 5
  Week 24: number analyzed (Participants) | 179 | 172
  Week 24 | 0 | 0
  Week 30: number analyzed (Participants) | 171 | 161
  Week 30 | 2 | 0
  Week 36: number analyzed (Participants) | 169 | 159
  Week 36 | 0 | 0
  Week 48: number analyzed (Participants) | 166 | 154
  Week 48 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit up to approximately 1.5 years.
Description: AE additional description
Groups:
- Treatment Period 1 TP1 SAF GP2015: Treatment Period 1 TP1 SAF GP2015
- Treatment Period 1 TP1 SAF Enbrel: Treatment Period 1 TP1 SAF Enbrel
- Treatment Period 2 TP2 SAF Continued GP2015: Treatment Period 2 TP2 SAF Continued GP2015
- Treatment Period 2 TP2 SAF Enbrel Switched to GP2015: Treatment Period 2 TP2 SAF Enbrel switched to GP2015
- Entire Study SAF GP2015: Entire study SAF GP2015
- Entire Study SAF Enbrel/GP2015: Entire study SAF Enbrel/GP2015
Arm/Group | Treatment Period 1 TP1 SAF GP2015 | Treatment Period 1 TP1 SAF Enbrel | Treatment Period 2 TP2 SAF Continued GP2015 | Treatment Period 2 TP2 SAF Enbrel Switched to GP2015 | Entire Study SAF GP2015 | Entire Study SAF Enbrel/GP2015
All-Cause Mortality (participants affected / at risk) | 0/186 | 1/190 | 0/175 | 0/166 | 0/186 | 1/190
Serious Adverse Events (participants affected / at risk) | 1/186 | 5/190 | 4/175 | 4/166 | 5/186 | 9/190
Other Adverse Events (participants affected / at risk) | 52/186 | 64/190 | 42/175 | 37/166 | 79/186 | 81/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1 TP1 SAF GP2015 (N=186) | Treatment Period 1 TP1 SAF Enbrel (N=190) | Treatment Period 2 TP2 SAF Continued GP2015 (N=175) | Treatment Period 2 TP2 SAF Enbrel Switched to GP2015 (N=166) | Entire Study SAF GP2015 (N=186) | Entire Study SAF Enbrel/GP2015 (N=190)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Salivary gland cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1 TP1 SAF GP2015 (N=186) | Treatment Period 1 TP1 SAF Enbrel (N=190) | Treatment Period 2 TP2 SAF Continued GP2015 (N=175) | Treatment Period 2 TP2 SAF Enbrel Switched to GP2015 (N=166) | Entire Study SAF GP2015 (N=186) | Entire Study SAF Enbrel/GP2015 (N=190)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 1 | 2 | 4 | 6
Injection site reaction (General disorders) | 13 | 35 | 0 | 6 | 13 | 37
Bronchitis (Infections and infestations) | 2 | 4 | 2 | 2 | 4 | 6
Cystitis (Infections and infestations) | 2 | 4 | 2 | 1 | 4 | 5
Nasopharyngitis (Infections and infestations) | 9 | 4 | 13 | 9 | 18 | 12
Pharyngitis (Infections and infestations) | 1 | 3 | 2 | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 9 | 9 | 13 | 15
Urinary tract infection (Infections and infestations) | 8 | 8 | 7 | 2 | 13 | 8
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 2 | 4 | 2
Alanine aminotransferase increased (Investigations) | 8 | 4 | 4 | 6 | 12 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 3 | 0 | 8 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 4 | 1 | 5
Hypertension (Vascular disorders) | 2 | 2 | 2 | 0 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Terms related to publication are part of the contract templates between Sponsor and sites/investigators. In general, these terms outlined that authorship of any publications relating to the clinical study shall be determined by agreement with the Sponsor. Sponsor reserves the right to request amendments or deletions to proposed publications, or request that any publication or presentation be delayed up to four months. A very limited number of exceptions can be granted to modify these terms.